CLINICAL TRIAL: NCT04014140
Title: Long-term Graft Patency Outcomes of LIMA-LAD Post-CABG Surgery Based on iFR Measurements.
Brief Title: iFR Guided Coronary Artery Bypass Grafting Surgery
Acronym: iCABG
Status: Recruiting | Type: Observational
Sponsor: Prakash Punjabi (Other)
Responsible Party: Sponsor-Investigator, Prakash Punjabi, Consultant Cardiothoracic Surgeon, Imperial College Healthcare NHS Trust
Organization: Imperial College Healthcare NHS Trust (Other)
Other Study IDs: 17HH3875
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Ischaemic Heart Disease; Coronary Artery Disease; Coronary Stenosis
Keywords: Instantaneous wave-free ratio (iFR); Coronary Artery Bypass Grafting (CABG)
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multi-vessel coronary artery disease (MVCAD): iFR measurements will be taken pre-operatively during the invasive coronary angiography.
  Interventions: Procedure: Coronary artery bypass grafting surgery (CABG)

INTERVENTIONS:
Procedure: Coronary artery bypass grafting surgery (CABG) — Patients with MVCAD will undergo CABG as per standard of care.

SUMMARY:
The expected outcome of better and improved patency of bypass grafts and its direct relation to pre-operative iFR measurements of stenosis as compared to direct visual physiology of stenosis in the coronary angiogram.

To establish the correlation between the use of intracoronary physiology and improved graft patency at 12 months for patients undergoing CABG surgery.

It is a minimum of 28 and a maximum of 100 patients single-centre proof or concept/ observational study/ pilot study.

DETAILED DESCRIPTION:
Patients suffering from coronary artery disease undergo coronary artery bypass grafting surgery (CABG) as the standard of care. The selection of which vessels to bypass is usually at the discretion of the surgeon forming an opinion based on the pre-operative angiographic imaging. Intra-coronary physiology (iFR measurements) is more accurate to determine the level of damage to the coronary arteries; however, currently it is not used for CABG pre-assessment, but only for percutaneous intervention also known as stenting as it has been shown to improve outcomes. Although, the use of intracoronary physiology has not been extensively studied or validated in patients undergoing CABG.

Patients with multi-vessel coronary artery disease (CAD) who are planned for surgical revascularization with coronary artery bypass grafting (CABG), will have iFR measurement taken during invasive coronary angiography as part of standard care, they will undergo CABG and will have echocardiography at 3 months and computed tomography coronary angiography (CTCA) at 12 months.

Early graft failure will be assessed by the presentation of any clinical symptoms, major adverse cardiovascular and cerebrovascular events (MACCE) and echocardiography at 3 months. The endpoint will be graft patency as assessed by CT coronary angiography at 12 months.

Anticipated recruitment is 12-24 months. Follow-up with echocardiography at 3 months and a CTCA at 12 months. Quality of Life questionnaire will be completed by the patient at 3 and 12 months during the follow-up appointment.

Patients will continue on optimal medical therapy. Clinic visit and quality of life scale questionnaires will be recorded at 3 and 12 months and echocardiography will be assessed at 3 months. Graft patency at 12 months will be assessed with a CT coronary angiography.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age of 25 to 80 years of age
2. Willing to participate and able to understand, read and sign the informed consent form (ICF) before standard of care elective CABG surgery
3. Undergoing isolated first-time elective CABG surgery
4. Available pre-operative angiography data with iFR measurements done during the pre-operative angiography

EXCLUSION CRITERIA

1. Emergency CABG surgery
2. Ejection Fraction≤ 40%
3. Severe valvular heart disease

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort study - approximately 250 pts Prospective cohort study - minimum 28 pts - maximum 100 pts
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Graft patency | 12 months
  The primary endpoint will be graft patency as assessed by CT coronary angiography at 12 months.

SECONDARY OUTCOMES:
Quality of Life Questionnaire | 3 and 12 months
  Patient's view in their quality of life
Composite of MACE (MI, Death, stroke, repeat revascularisation) | 12 months
  Assessed by the presentation of clinical symptoms and echocardiography during a follow-up visit at 3 months or anytime within 12 months.
Any episode of reintervention | 12 months
  Patient undergoing repeat reintervention
Incidence of Myocardial infarction | 12 months
  Assessed by the presentation of clinical symptoms, echocardiography during a follow-up visit at 3 months or anytime within 12 months and in addition, evidence of percutaneous or surgical revascularisation within the last 12 months.
Incidence of Stroke | 12 months
  Assessed by the presentation of clinical symptoms during a follow-up visit at 3 and 12 months or anytime within 12 months.
Left ventricular function at 3 months with an echocardiography | 3 months
  Cardiac functional assessment at 3 months post-opereatively
Incidence of Death (all-cause) | 12 months
  Patient deceased
Incident of Death (cardiovascular) | 12 months
  Patient deceased

CONTACTS AND LOCATIONS:
Overall Officials: Prakash P Punjabi, MBBS,MCh,FRCS,FFST,FESC,FCCP, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust - Hammersmith Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 36 months
Access Criteria: According to study protocol